CLINICAL TRIAL: NCT02850367
Title: The Effect of NO Precursors on Physiological Responses to Exercise
Brief Title: Effect of NO Precursors on Physiological Responses to Exercise
Acronym: NO-SUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 38RC14.430
Record Dates: First submitted 2016-05-18; First posted 2016-08-01 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Physiology
MeSH Terms: interventions — Nitrates; Arginine; Citrulline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acute intake (Active Comparator): Evaluation after acute intake of the food supplement.
  Interventions: Dietary Supplement: Nitrate; Dietary Supplement: Nitrate and L-Arginine; Dietary Supplement: Nitrate and L-Citrulline; Dietary Supplement: Placebo; Biological: Evaluation of post-ischemic vascular reactivity; Biological: Neuromuscular evaluations
- Chronic intake (Active Comparator): Evaluation before and after chronic intake of the food supplement.
  Interventions: Dietary Supplement: Nitrate and L-Citrulline; Dietary Supplement: Placebo; Biological: Evaluation of post-ischemic vascular reactivity; Biological: Neuromuscular evaluations

INTERVENTIONS:
Dietary Supplement: Nitrate — Subjects will be supplemented orally either acutely or chronically (4-8 weeks) with NO precursors.
  Arms: Acute intake
Dietary Supplement: Nitrate and L-Arginine — Subjects will be supplemented orally either acutely or chronically (4-8 weeks) with NO precursors.
  Arms: Acute intake
Dietary Supplement: Nitrate and L-Citrulline — Subjects will be supplemented orally either acutely or chronically (4-8 weeks) with NO precursors.
Dietary Supplement: Placebo — Subjects will be supplemented orally either acutely or chronically (4-8 weeks) with a placebo.
Biological: Evaluation of post-ischemic vascular reactivity — After the intake of the supplement. Concentration of hemoglobin (g/mL) in the quadriceps with the device : NIRS system Oxymon, ARTINIS.
Biological: Neuromuscular evaluations — After the intake of the supplement. Measure the stretching force in the ankle (N)

SUMMARY:
NO is an ubiquitous molecule contributing to many physiological functions such as vasodilation, immune and oxidative stress responses. NO production can be supplemented either by providing substrate to the NO-synthase (L-Arginine and L-Citruline) or by providing nitrate which can lead to NO. In the present project the investigators evaluate the effect of various acute and chronic oral NO precursors supplementation on exercise performance and responses in healthy young and older subjects.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary subjects
* No cardiovascular, respiratory, metabolic and neurological disorders

Exclusion Criteria:

* Body mass index > 28 kg.m-2
* Smoker
* Alcool intake > 10g/day
* Psychiatric diseases
* Subjects under treatment able to interfere with their cardiovascular, metabolic and neurological status

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Neuromuscular evaluations | 3 half days
  After the intake of the supplement. Measure the stretching force in the ankle (N)
Evaluation of post-ischemic vascular reactivity | 3 half days
  After the intake of the supplement. Concentration of hemoglobin (g/mL) in the quadriceps with the device : NIRS system Oxymon, ARTINIS.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Doutreleau, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones AM. Dietary nitrate supplementation and exercise performance. Sports Med. 2014 May;44 Suppl 1(Suppl 1):S35-45. doi: 10.1007/s40279-014-0149-y. PMID 24791915
- [Background] Kapil V, Weitzberg E, Lundberg JO, Ahluwalia A. Clinical evidence demonstrating the utility of inorganic nitrate in cardiovascular health. Nitric Oxide. 2014 Apr 30;38:45-57. doi: 10.1016/j.niox.2014.03.162. Epub 2014 Mar 18. PMID 24650698
- [Background] Kelly J, Vanhatalo A, Wilkerson DP, Wylie LJ, Jones AM. Effects of nitrate on the power-duration relationship for severe-intensity exercise. Med Sci Sports Exerc. 2013 Sep;45(9):1798-806. doi: 10.1249/MSS.0b013e31828e885c. PMID 23475164
- [Background] Lasker GF, Matt CJ, Badejo AM Jr, Casey DB, Dhaliwal JS, Murthy SN, Kadowitz PJ. Intracavernosal administration of sodium nitrite as an erectile pharmacotherapy. Can J Physiol Pharmacol. 2010 Jul;88(7):770-6. doi: 10.1139/y10-032. PMID 20651825
- [Background] Lee M, Gandevia SC, Carroll TJ. Cortical voluntary activation can be reliably measured in human wrist extensors using transcranial magnetic stimulation. Clin Neurophysiol. 2008 May;119(5):1130-8. doi: 10.1016/j.clinph.2007.12.018. Epub 2008 Mar 4. PMID 18308630
- [Background] Liu TH, Wu CL, Chiang CW, Lo YW, Tseng HF, Chang CK. No effect of short-term arginine supplementation on nitric oxide production, metabolism and performance in intermittent exercise in athletes. J Nutr Biochem. 2009 Jun;20(6):462-8. doi: 10.1016/j.jnutbio.2008.05.005. Epub 2008 Aug 15. PMID 18708287
- [Background] Martin MJ, Jimenez MD, Motilva V. New issues about nitric oxide and its effects on the gastrointestinal tract. Curr Pharm Des. 2001 Jul;7(10):881-908. doi: 10.2174/1381612013397645. PMID 11472246
- [Background] Moinard C, Nicolis I, Neveux N, Darquy S, Benazeth S, Cynober L. Dose-ranging effects of citrulline administration on plasma amino acids and hormonal patterns in healthy subjects: the Citrudose pharmacokinetic study. Br J Nutr. 2008 Apr;99(4):855-62. doi: 10.1017/S0007114507841110. Epub 2007 Oct 22. PMID 17953788
- [Background] Moncada S. The L-arginine: nitric oxide pathway, cellular transduction and immunological roles. Adv Second Messenger Phosphoprotein Res. 1993;28:97-9. No abstract available. PMID 8398422
- [Background] Moncada S, Higgs A. The L-arginine-nitric oxide pathway. N Engl J Med. 1993 Dec 30;329(27):2002-12. doi: 10.1056/NEJM199312303292706. No abstract available. PMID 7504210
- [Background] Morris CR, Morris SM Jr, Hagar W, Van Warmerdam J, Claster S, Kepka-Lenhart D, Machado L, Kuypers FA, Vichinsky EP. Arginine therapy: a new treatment for pulmonary hypertension in sickle cell disease? Am J Respir Crit Care Med. 2003 Jul 1;168(1):63-9. doi: 10.1164/rccm.200208-967OC. Epub 2003 Mar 5. PMID 12626350
- [Background] Ochiai M, Hayashi T, Morita M, Ina K, Maeda M, Watanabe F, Morishita K. Short-term effects of L-citrulline supplementation on arterial stiffness in middle-aged men. Int J Cardiol. 2012 Mar 8;155(2):257-61. doi: 10.1016/j.ijcard.2010.10.004. Epub 2010 Nov 9. PMID 21067832
- [Background] Park JW, Piknova B, Kurtz J, Seetharaman S, Wagner SJ, Schechter AN. Effect of storage on levels of nitric oxide metabolites in platelet preparations. Transfusion. 2013 Mar;53(3):637-44. doi: 10.1111/j.1537-2995.2012.03777.x. Epub 2012 Jul 15. PMID 22804724
- [Background] Pavy B, Iliou MC, Meurin P, Tabet JY, Corone S; Functional Evaluation and Cardiac Rehabilitation Working Group of the French Society of Cardiology. Safety of exercise training for cardiac patients: results of the French registry of complications during cardiac rehabilitation. Arch Intern Med. 2006 Nov 27;166(21):2329-34. doi: 10.1001/archinte.166.21.2329. PMID 17130385
- [Background] Peacock O, Tjonna AE, James P, Wisloff U, Welde B, Bohlke N, Smith A, Stokes K, Cook C, Sandbakk O. Dietary nitrate does not enhance running performance in elite cross-country skiers. Med Sci Sports Exerc. 2012 Nov;44(11):2213-9. doi: 10.1249/MSS.0b013e3182640f48. PMID 22874535
- [Background] Perrey S. Non-invasive NIR spectroscopy of human brain function during exercise. Methods. 2008 Aug;45(4):289-99. doi: 10.1016/j.ymeth.2008.04.005. Epub 2008 Jun 6. PMID 18539160
- [Background] Preli RB, Klein KP, Herrington DM. Vascular effects of dietary L-arginine supplementation. Atherosclerosis. 2002 May;162(1):1-15. doi: 10.1016/s0021-9150(01)00717-1. PMID 11947892
- [Background] Rupp T, Esteve F, Bouzat P, Lundby C, Perrey S, Levy P, Robach P, Verges S. Cerebral hemodynamic and ventilatory responses to hypoxia, hypercapnia, and hypocapnia during 5 days at 4,350 m. J Cereb Blood Flow Metab. 2014 Jan;34(1):52-60. doi: 10.1038/jcbfm.2013.167. Epub 2013 Sep 25. PMID 24064493
- [Background] Rupp T, Leti T, Jubeau M, Millet GY, Bricout VA, Levy P, Wuyam B, Perrey S, Verges S. Tissue deoxygenation kinetics induced by prolonged hypoxic exposure in healthy humans at rest. J Biomed Opt. 2013 Sep;18(9):095002. doi: 10.1117/1.JBO.18.9.095002. PMID 24064948
- [Background] Rupp T, Jubeau M, Millet GY, Wuyam B, Levy P, Verges S, Perrey S. Muscle, prefrontal, and motor cortex oxygenation profiles during prolonged fatiguing exercise. Adv Exp Med Biol. 2013;789:149-155. doi: 10.1007/978-1-4614-7411-1_21. PMID 23852489
- [Background] Rupp T, Jubeau M, Wuyam B, Perrey S, Levy P, Millet GY, Verges S. Time-dependent effect of acute hypoxia on corticospinal excitability in healthy humans. J Neurophysiol. 2012 Sep;108(5):1270-7. doi: 10.1152/jn.01162.2011. Epub 2012 Jun 13. PMID 22696539
- [Background] Rupp T, Perrey S. Effect of severe hypoxia on prefrontal cortex and muscle oxygenation responses at rest and during exhaustive exercise. Adv Exp Med Biol. 2009;645:329-34. doi: 10.1007/978-0-387-85998-9_49. PMID 19227490
- [Background] Sidhu SK, Bentley DJ, Carroll TJ. Locomotor exercise induces long-lasting impairments in the capacity of the human motor cortex to voluntarily activate knee extensor muscles. J Appl Physiol (1985). 2009 Feb;106(2):556-65. doi: 10.1152/japplphysiol.90911.2008. Epub 2008 Dec 4. PMID 19056999
- [Background] Siervo M, Lara J, Ogbonmwan I, Mathers JC. Inorganic nitrate and beetroot juice supplementation reduces blood pressure in adults: a systematic review and meta-analysis. J Nutr. 2013 Jun;143(6):818-26. doi: 10.3945/jn.112.170233. Epub 2013 Apr 17. PMID 23596162
- [Background] Sunderland KL, Greer F, Morales J. VO2max and ventilatory threshold of trained cyclists are not affected by 28-day L-arginine supplementation. J Strength Cond Res. 2011 Mar;25(3):833-7. doi: 10.1519/JSC.0b013e3181c6a14d. PMID 20581700
- [Background] Takeda K, Machida M, Kohara A, Omi N, Takemasa T. Effects of citrulline supplementation on fatigue and exercise performance in mice. J Nutr Sci Vitaminol (Tokyo). 2011;57(3):246-50. doi: 10.3177/jnsv.57.246. PMID 21908948
- [Background] Tang JE, Lysecki PJ, Manolakos JJ, MacDonald MJ, Tarnopolsky MA, Phillips SM. Bolus arginine supplementation affects neither muscle blood flow nor muscle protein synthesis in young men at rest or after resistance exercise. J Nutr. 2011 Feb;141(2):195-200. doi: 10.3945/jn.110.130138. Epub 2010 Dec 29. PMID 21191143
- [Background] Vanhatalo A, Bailey SJ, DiMenna FJ, Blackwell JR, Wallis GA, Jones AM. No effect of acute L-arginine supplementation on O(2) cost or exercise tolerance. Eur J Appl Physiol. 2013 Jul;113(7):1805-19. doi: 10.1007/s00421-013-2593-z. Epub 2013 Feb 20. PMID 23423302
- [Background] Vega-Villa K, Pluta R, Lonser R, Woo S. Quantitative Systems Pharmacology Model of NO Metabolome and Methemoglobin Following Long-Term Infusion of Sodium Nitrite in Humans. CPT Pharmacometrics Syst Pharmacol. 2013 Jul 31;2(7):e60. doi: 10.1038/psp.2013.35. PMID 23903463
- [Background] Verges S, Maffiuletti NA, Kerherve H, Decorte N, Wuyam B, Millet GY. Comparison of electrical and magnetic stimulations to assess quadriceps muscle function. J Appl Physiol (1985). 2009 Feb;106(2):701-10. doi: 10.1152/japplphysiol.01051.2007. Epub 2008 Aug 28. PMID 18756009
- [Background] Villanueva C, Giulivi C. Subcellular and cellular locations of nitric oxide synthase isoforms as determinants of health and disease. Free Radic Biol Med. 2010 Aug 1;49(3):307-16. doi: 10.1016/j.freeradbiomed.2010.04.004. Epub 2010 Apr 11. PMID 20388537
- [Background] Vuillemin A, Oppert JM, Guillemin F, Essermeant L, Fontvieille AM, Galan P, Kriska AM, Hercberg S. Self-administered questionnaire compared with interview to assess past-year physical activity. Med Sci Sports Exerc. 2000 Jun;32(6):1119-24. doi: 10.1097/00005768-200006000-00013. PMID 10862539
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Wylie LJ, Kelly J, Bailey SJ, Blackwell JR, Skiba PF, Winyard PG, Jeukendrup AE, Vanhatalo A, Jones AM. Beetroot juice and exercise: pharmacodynamic and dose-response relationships. J Appl Physiol (1985). 2013 Aug 1;115(3):325-36. doi: 10.1152/japplphysiol.00372.2013. Epub 2013 May 2. PMID 23640589
- [Background] Wylie LJ, Mohr M, Krustrup P, Jackman SR, Ermiotadis G, Kelly J, Black MI, Bailey SJ, Vanhatalo A, Jones AM. Dietary nitrate supplementation improves team sport-specific intense intermittent exercise performance. Eur J Appl Physiol. 2013 Jul;113(7):1673-84. doi: 10.1007/s00421-013-2589-8. Epub 2013 Feb 1. PMID 23370859
- [Background] Zhu Q, Yue X, Tian QY, Saren G, Wu MH, Zhang Y, Liu TT. Effect of L-arginine supplementation on blood pressure in pregnant women: a meta-analysis of placebo-controlled trials. Hypertens Pregnancy. 2013;32(1):32-41. doi: 10.3109/10641955.2012.697952. Epub 2012 Sep 7. PMID 22957482
- [Result] LE Roux-Mallouf T, Vallejo A, Pelen F, Halimaoui I, Doutreleau S, Verges S. Synergetic Effect of NO Precursor Supplementation and Exercise Training. Med Sci Sports Exerc. 2020 Nov;52(11):2437-2447. doi: 10.1249/MSS.0000000000002387. PMID 33064413